CLINICAL TRIAL: NCT02391181
Title: An Open-label, Randomized, Crossover-design Bioequivalence Study With Pharmacokinetic Endpoints, Comparing a Single Dose of Iron Sucrose Azad Injection of Azad Pharma Corporation (AG), With a Single Dose of Venofer® Injection of Vifor Corporation (AG) in Healthy Adult Volunteers Under Fasting Conditions
Brief Title: Bioequivalence Study With Pharmacokinetic Endpoints, Comparing a Single Dose of Iron Sucrose Azad Injection of Azad Pharma Corporation (AG), With a Single Dose of Venofer® Injection of Vifor Corporation (AG) in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Azad Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AZAD-BE01
Record Dates: First submitted 2015-01-22; First posted 2015-03-18 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Healthy Volunteers
Keywords: Bioequivalence; Iron Status
MeSH Terms: interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- test product (Experimental): Iron sucrose injection solution 100mg (5 mL single dose ampoule 20mg/mL elemental iron as iron sucrose in water for injection)
  Interventions: Drug: Iron Sucrose Azad
- reference product (Active Comparator): Iron sucrose injection solution 100mg (5 mL single dose vial 20mg/mL elemental iron as iron sucrose in water for injection)
  Interventions: Drug: Venofer®

INTERVENTIONS:
Drug: Iron Sucrose Azad — Test product Iron Sucrose Azad will be administered intravenously via a 18 gauge (18G) needle. For intravenous injection, a 5 mL single dose of test product (each mL containing 20 mg/mL elemental iron as iron sucrose in water for injection) will be diluted in 0.9% isotonic sterile sodium chloride (NaCl) up to 15 mL. The injection solution will be intravenously administered to the forearm vein, resulting in a total injection volume of 15 mL administered over a period of 5 minutes.
  Arms: test product
Drug: Venofer® — Reference product Venofer® will be administered intravenously via a 18 gauge (18G) needle. For intravenous injection, a 5 mL single dose of reference product (each mL containing 20 mg/mL elemental iron as iron sucrose in water for injection) will be diluted in 0.9% isotonic sterile sodium chloride (NaCl) up to 15 mL. The injection solution will be intravenously administered to the forearm vein, resulting in a total injection volume of 15 mL administered over a period of 5 minutes.
  Arms: reference product

SUMMARY:
A Clinical Trial to Demonstrate the Comparability of the Two Iron Sucrose Injection Solutions Iron Sucrose Azad of Azad Pharma AG and Venofer® of Vifor Pharma AG. The Hypothesis is That Both Iron Sucrose Injection Solutions Reveal the Same Active Substance Availability in the Blood Circuit.

DETAILED DESCRIPTION:
A single dose 100mg Iron Sucrose Azad (5 mL single dose vial, each mL containing 20 mg/mL elemental iron as iron sucrose in water for injection) of Azad Pharma AG or a single dose 100mg Venofer® (5 mL single dose vial, iron sucrose injection, United States Pharmacopeia (USP), 20 mg/mL) will be administered to healthy adult volunteers in a crossover-design. The assignment to either test or reference product in the crossover design is based on a randomization schedule. A wash-out period of at least 5 half-lives of iron sucrose was calculated in this crossover design which accounts an overall study duration of at least 10 days (max 19 days) for each volunteer. Overall the study participant has to attend the clinical site for 5 active study days.

The study follows the recommended format outlined 2013 by the European Medicines Agency (EMA), i.e. single-dose with primary variables being AUC and Cmax of baseline corrected total- and transferrin-bound serum iron. In addition baseline non-corrected values will be analysed due to the known variability in baseline iron levels (both intra- and inter-individual).

The assays for total- and transferrin-bound serum iron will be validated, in order to ensure dependable readouts as recommended by EMA.

ELIGIBILITY:
Inclusion Criteria:

* Male and female healthy volunteers within the age range of 18 to 45 years (both inclusive)
* Comprehension of the nature and purpose of the study and willingness to comply with the requirements of the entire procedure
* Subjects of good health based on previous medical history, physical examination, vital signs, electrocardiogram (ECG), and clinical laboratory tests assessed at the time of screening.
* Ferritin levels ≥ 30 µg/l for female and male subjects
* Transferrin ≥ 200 mg/dl for female and male subjects
* Hemoglobin levels ≥ 12 g/dl for female subjects and ≥ 13.5 g/dl for male subjects
* Females of childbearing potential must provide a negative urine pregnancy test at time of screening and have to be compliant with effective hormonal form of birth control throughout the whole study

Exclusion Criteria:

* Subjects with a BMI of < 19 kg/m2 and > 30 kg/m2
* Pregnancy (as determined by a positive urine pregnancy test at the screening or prior each crossover phase) or breast feeding
* Females with history of hypermenorrhea or menorrhagia
* Females with history of myoma, endometriosis or uterus hypoplasia or any other gynecological disorder
* History of iron deficiency within six months prior screening
* History of anemia within 1 year prior screening
* Presence of iron overload or disturbances in utilization of iron
* History or evidence of allergy or hypersensitivity to the active substance Iron Sucrose of both test and reference product, the finished test and reference product or any of its excipients (water for injection, sodium hydroxide)
* Hypersensitivity to other parenteral iron products
* Use of iron supplements or iron containing herbal or nutritional supplements within last three months prior to start of the study
* History of difficulty with donating blood or difficulty in accessibility of veins in left and right arm
* Donation of blood (one unit or 350 mL) within last three months prior first dose administration of the study drug
* Evidence of an active or suspected cancer, or a history of malignancy within the last 2 years, with the exception of patients with basal cell carcinoma that has been excised and cured
* History of any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) 6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study
* History of bleeding disorders or anticoagulant use
* History or other evidence of chronic pulmonary or cardiovascular disease associated with functional limitation
* History of uncontrolled severe seizure disorder.
* Any signs of acute infection or inflammation.
* History or other evidence of severe illness, or any other condition which would make the subject in the opinion of the investigator, unsuitable for the study
* Any clinically significant abnormal laboratory values on the laboratory evaluations, medical history or physical examination at the screening
* Positive Human Immunodeficiency Virus (HIV)/ Hepatitis B Virus (HBV)/ hepatitis C virus (HCV) serology tests at the time of the screening visit
* Abnormal 12-lead ECG at the time of screening that is considered to be clinically significant
* History or presence of severe or medical treated allergies or immune or inflammatory conditions (eg. systemic lupus erythematosus, rheumatoid arthritis)
* History of atopic allergy associated with severe asthma
* Recent history or ongoing kidney or liver dysfunction
* Any other major illness in last three months or any significant ongoing chronic medical illness
* Subjects who regularly use more than 2 units of alcohol per day (one unit of alcohol equals ½ liter of beer, 200mL wine or 50mL of spirits)or there is evidence of Cocaine, Amphetamines, Metformin, Tetrahydrocannabinol (THC), Methadone, 3,4-Methylendioxy-N-Methylamphetamin (MDMA), Morphine, Barbiturates, Benzodiazepines and Tricyclic antidepressants in urine at the screening)
* Heavy smokers (> 10 cigarettes/day) in the last three months prior to start of the study
* Any concomitant medication (except paracetamol and contraceptives) within the last two weeks, including over-the-counter and herbal products, prior to receiving the dose of study medication
* Participation in any clinical trial within last one months
* Subjects who are considered by the investigator to be non-compliant or unlikely to complete the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Comparative assessment of peak plasma concentration (Cmax) of baseline corrected total serum iron and serum transferrin-bound iron after administration of test and reference product. | -24.00, -12.00, -3.00 hours, at pre-dose (within 15 minutes prior to dosing), at 2, 5, 10, 15, 20, 30, 45 minutes and at 1.00, 1.30, 2.00, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 24.00 hours post-dose.
Comparative assessment of the area under the plasma concentration versus time curve (AUC) of baseline corrected total serum iron and serum transferrin-bound iron after administration of test and reference product. | -24.00, -12.00, -3.00 hours, at pre-dose (within 15 minutes prior to dosing), at 2, 5, 10, 15, 20, 30, 45 minutes and at 1.00, 1.30, 2.00, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 24.00 hours post-dose.

SECONDARY OUTCOMES:
Comparative assessment of peak plasma concentration (Cmax) of non-baseline corrected total serum iron and serum transferrin-bound iron after administration of test and reference product. | -24.00, -12.00, -3.00 hours, at pre-dose (within 15 minutes prior to dosing), at 2, 5, 10, 15, 20, 30, 45 minutes and at 1.00, 1.30, 2.00, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 24.00 hours post-dose.
Comparative assessment of the area under the plasma concentration versus time curve (AUC) of non-baseline corrected total serum iron and serum transferrin-bound iron after administration of test and reference product. | -24.00, -12.00, -3.00 hours, at pre-dose (within 15 minutes prior to dosing), at 2, 5, 10, 15, 20, 30, 45 minutes and at 1.00, 1.30, 2.00, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 24.00 hours post-dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria